CLINICAL TRIAL: NCT04286763
Title: Factors Influencing Occurence Of Hight Level of Biliary Stricture Due to Operative Bile Duct Injury
Brief Title: Factors Influencing Occurrence Of Hilar Biliary Stricture In Case of Bile Duct Injury
Status: Completed | Type: Observational
Sponsor: University of Oran 1 (Other)
Responsible Party: Principal Investigator, Anisse Tidjane, Ph.D, University of Oran 1
Other Study IDs: UOran1bileductinjury
Record Dates: First submitted 2020-02-20; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Bile Duct Injury
Keywords: bile duct injury; surgery; laparoscopy; cholecystectomy; Bile duct stricture
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hilar stricture: Bile duct Stricture (corresponding to E3, E4 and E5 from of Strasberg. -According to the classification proposed by Strasberg of operative bile duct injuries).
  Interventions: Diagnostic Test: Biliary RMI and CT scan.
- Low level Stricture: Bile duct Stricture (corresponding to E1 and E2 from Strasberg. -According to the classification proposed by Strasberg of operative bile duct injuries).
  Interventions: Diagnostic Test: Biliary RMI and CT scan.

INTERVENTIONS:
Diagnostic Test: Biliary RMI and CT scan. — For a good appreciation of the anatomy of the biliary lesion, an MRI was systematically performed on all our patients.
  For a good appreciation of the presence of an associated vascular lesion, a CT-scan was systematically performed on all our patients.

SUMMARY:
The bile duct injury is a complication that occurs mainly after the cholecystectomy. Bile duct stricture is one of complications of this unwitting iatrogenic injury, the outcomes of surgery in this case are worse when the level of the stricture is above the helium.

So what are factors influencing the occurrence of this high level bile duct obstruction ?

DETAILED DESCRIPTION:
The objective of this study was to answer a simple question, what are the factors influencing the occurrence of high level -called hilar biliary stricture? To answer this question, a retrospective study was carried out on the files of patients operated for biliary stenosis after operative trauma of the bile ducts in our department over a period from January 2010 to May 2018. Only patients operated in biliary stricture (Grade E Strasberg) was included.

A univariate and muntivariate logistic regression analysis was performed to determine the factors influencing the occurrence of hilar stenosis. data entry and analysis was done using SPSS V20.0 software.

ELIGIBILITY:
Inclusion Criteria:

* all cases with biliary stricture following an operative bile duct injury.

Exclusion Criteria:

* cases of biliary stricture following an non operative bile duct injury (Blind or penetrating abdominal trauma , radiological or endoscopic maneuvers).
* cases of biliary stricture following hepatectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of biliary structure admitted for the management of an operative bile duct injury in the hepatobiliary surgery and liver transplant department of EHU-1st November 1954 / Oran, Algeria.
  No geographic origin is excluded, patients are admitted in our department following a meducal consultation, a medical orientation or an emergency evacuation.
  Any patient meeting the inclusion criteria is eligible for this study after informed consent concerning the use of their personal data for research purposes with respect for anonymity and professional secrecy.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Factors influencing occurrence of hilar stricture (E3,E4,E5) | from the date of the surgery that caused the biliary injury to the date of transfer to our structure for treatment. in our series, the period varies from 8 weeks to 10 years after the occurrence of operative bile duct injury during initial surgery.
  all the variables related to the patient, his disease and the course of the surgical intervention which caused the biliary trauma was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Noureddine Benmaarouf, Pr, Study Director — University of Oran 1
Locations (1):
- Tidjane Anisse, Oran, Algeria

IPD SHARING:
Plan to Share IPD: Undecided